CLINICAL TRIAL: NCT04434703
Title: Alveolar Ridge Preservation Following Tooth Extraction Using Advanced Platelet Rich Fibrin (A-PRF) Versus Platelet Rich Fibrin (PRF) A Randomized Clinical Trail :Comparative Study
Brief Title: Alveolar Ridge Preservation Following Tooth Extraction Using Advanced Platelet Rich Fibrin (A-PRF) Versus Platelet Rich Fibrin (PRF)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Reem Mahmoud AbdAlhameed AbuBasha, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 6-3-1
Record Dates: First submitted 2020-06-13; First posted 2020-06-17 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Alveolar Bone Resorption
MeSH Terms: interventions — Blood Coagulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Platelet rich fibrin (PRF) (Active Comparator): Platelet rich fibrin is the secoond generation of platelet concentrates which is an autogenous biomaterial that is prepared from the patient's own blood
  Interventions: Procedure: Platelet rich fibrin (PRF)
- Advanced platelet rich fibrin (A-PRF) (Experimental): Advanced platelet rich fibrin is the last modification of PRF which is expected to contain a relatively greater number of white blood cellsand growth factors
  Interventions: Procedure: Advanced platelet rich fibrin (A-PRF)
- blood clot (Placebo Comparator): normal healing of the wound without adding any biomaterial
  Interventions: Procedure: blood clot

INTERVENTIONS:
Procedure: Platelet rich fibrin (PRF) — following atraumatic extraction of the tooth using periotomes , 10 ml of patient's blood will be drawn by vein puncture of the antecubital vein and prepared in a centrifuge at 3000 rpm for 10 minutes then criss horizontal mattress suture will be applied to close the extraction wound
  Arms: Platelet rich fibrin (PRF)
Procedure: Advanced platelet rich fibrin (A-PRF) — following atraumatic extraction of the tooth using periotomes , 10 ml of patient's blood will be drawn by vein puncture of the antecubital vein and prepared in a centrifuge at 1300 rpm for 8 minutes then criss horizontal mattress suture will be applied to close the extraction wound
  Arms: Advanced platelet rich fibrin (A-PRF)
Procedure: blood clot — following atraumatic extraction of the tooth using periotomes, no bio-addative will be added and criss horizontal mattress suture will be applied to close the extraction wound
  Arms: blood clot

SUMMARY:
the aim of this study is clinically and radiographically evaluate the use of advance platelet rich fibrin (A-PRF) versus platelet rich fibrin (PRF) in preservation of alveolar ridge following tooth extraction

DETAILED DESCRIPTION:
systemically healthy patients who have at least one non-restorable tooth in the upper inter-bicuspid region and are not seeking immediate or early implant treatment will be allocated in this study after performing nonsurgical periodontal therapy and preoperative periapical therapy to evaluate and improve the condition of the periodontal tissues.

Anesthesia will be given then flapless atraumatic extraction using periotomes followed by forceps after luxation. For all groups, the socket will be debrided using curette then

* group A, the socket will be filled with A.PRF
* group B the socket will be filled with PRF.
* group C no bio-additive will be added.
* Criss cross horizontal mattress suture will be applied to close the extraction wound.

PRF and A-PRF preparation :

10 ml of blood will be drawn from each patient by vein puncture of the antecubital vein.

* Plateletr ich fibrin (PRF) is 3000 rpm and 10 minutes without addition of anticoagulant
* Advanced platelet rich fibrin (A-PRF) is 1300 rpm and 8 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with at least one non restorable tooth in upper inter-bicuspid region.
* Stable periodontal condition with no acute periapical infection.
* Systematically healthy conditions.
* Cooperative patients.
* Intact buccal plate of bone.

Exclusion Criteria:

* Smokers.
* Patients seeking immediate or early implants.
* Pregnant females.
* Bone diseases.
* Drugs and diseases that may affect platelet count or function.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-07-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in bucco-lingual dimensions | 6 months
  clinical measurement using bone caliper in mm numerical

SECONDARY OUTCOMES:
change in alveolar bone height | 6 months
  radiographic measurement using CBCT in mm numerical
bone dentistry | 6 months
  radiographic measurement using CBCT
soft tissue healing | 6 months
  clinical measurement using landr et al index (healing index) in numerical
postoperative pain scores | 2 weeks
  clinical measurement using VAS scale in numerical where No pain (0-4 mm) - mild pain (5-44 mm) -moderate pain (45-74 mm), and severe pain (75- 100 mm).

CONTACTS AND LOCATIONS:
Locations (1):
- School of dentistry , Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
it will include participant's contacts ( name, age , phone number , address ,medical and dental history , periodontal condition) ,periodontal chart and preoperative radiograph